CLINICAL TRIAL: NCT06447233
Title: An Exploratory Analysis of Patient Perspectives Regarding the Medicaid Title XIX Sterilization Consent Form
Brief Title: Patient Perspectives Medicaid Title XIX Sterilization Consent Form
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: AAAU9746
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Patient Satisfaction
Keywords: Sterilization; Coercion; Understanding; Satisfaction
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this survey and interview study is to learn about patient experience consenting for permanent contraception using the Medicaid Title XIX Sterilization Consent form. The main questions it aims to answer are:

* To explore patient perspectives on and understanding of the current consenting process for obtaining permanent contraception as it relates to the Medicaid Title XIX Sterilization consent form.
* To explore patient experience with the current consenting process, and thoughts regarding the ideal consenting process including how it would differ from the one currently in place, if at all.

Participants will complete a 10-15 minute survey and be offered participation in an in-depth one-on-one interview.

DETAILED DESCRIPTION:
The United States has a long history of coerced sterilization which was influenced by the eugenics and population control movements of the early and mid-20th century, respectively. The Medicaid Title XIX Sterilization Consent Form was created in response to these forced sterilizations to protect patients, but in recent years there have been questions regarding whether these forms are instead creating barriers to care for already marginalized populations. Prior studies demonstrated decreased rates of completion of postpartum permanent contraception requests secondary to invalid consent forms and negative attitudes among OBGYNs, including concerns regarding the ethics behind the forms. To date, there is very limited literature exploring patient perspectives. This will be a mixed methods study in which bilingual surveys will be distributed via REDCap to patients seeking permanent contraception at Columbia University affiliated OBGYN practices and complete in-depth interviews exploring patient experiences consenting for permanent contraception, and what an ideal consenting process might look like to them.

ELIGIBILITY:
Inclusion Criteria:

* Seeking permanent contraception procedure through a Columbia University practice
* English or Spanish speaking
* Completed the Medicaid Title XIX Consent Form

Exclusion Criteria:

-Currently pregnant and seeking immediate postpartum permanent contraception

Min Age: 21 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study participants will be patients seeking care at Columbia University affiliated OBGYN practices. The Columbia University affiliated OBGYN practices serve the Washington Heights and Inwood communities of New York City. The patient population is majority Hispanic and foreign-born. Approximately half of patients seeking permanent contraception are Spanish speaking.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient experience with the Medicaid Title XIX Sterilization consent form | Day 1, up to 1 hour
  Patient perspectives on and understanding of the current consenting process for obtaining permanent contraception as it relates to the Medicaid Title XIX Sterilization consent form. Patients' responses to interview questions will be translated into coded data using Dedoose, and grouped coded data will inform patterns of patient experience. Quantitative software will be used to analyze survey responses using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Levi, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States